CLINICAL TRIAL: NCT02368431
Title: Effectiveness of Zonisamide in the Treatment of Alcohol Dependent Veterans
Brief Title: Effectiveness of Zonisamide in Alcohol Dependent Veterans
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Funding ended prematurely
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLNA-003-14S; ICX001012A (Other: VA Connecticut Healthcare System)
Record Dates: First submitted 2015-02-14; First posted 2015-02-23 (Estimated); Results first posted 2020-06-02 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol Use Disorder; Alcoholism; Alcohol Dependence; Zonisamide; Alcoholic Intoxication; Drinking Behaviors; Anticonvulsants
MeSH Terms: conditions — Alcoholism; Alcoholic Intoxication; Drinking Behavior | interventions — Zonisamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Zonisamide (Experimental): Subjects will receive zonisamide titrated to a target dose of 500mg orally, daily, double-blind (Titration of dose to 500mg oral, daily, over 8 weeks, then 7 weeks of treatment at that dose). Subjects may increase their dose to 600mg daily during the target treatment period if it is thought to be beneficial.
  Interventions: Drug: Zonisamide
- Placebo (Placebo Comparator): Patients will receive placebo pills that are made to match the zonisamide medication (via over-encapsulation, double-blind, subjects will receive same number of capsules as the active medication group)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zonisamide — Titration of dose to 500mg oral, daily, over 8 weeks, then 7 weeks of treatment at that dose
  Other Names: Zonegran
  Arms: Zonisamide
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled, double-blind, 16 week trial of the medication zonisamide for the treatment of heavy drinking alcoholic Veterans.

DETAILED DESCRIPTION:
This is a 16-week randomized, double blind, placebo-controlled trial designed to determine the effectiveness of zonisamide treatment for reducing heavy drinking and overall drinking in 160 treatment-seeking, regularly heavy drinking, alcohol-dependent Veterans who want to quit drinking or reduce consumption to non-hazardous levels. The investigators will use state-of-the-art methodology and outcome assessments, including medical management (MM) therapy (a minimal behavioral intervention aimed at reinforcing treatment goals and adherence to medication), which is simple and easily implemented in primary care settings. The use of MM in the study will increase the generalizability of results, allowing a more accurate assessment of zonisamide's effectiveness than if a more intensive behavioral intervention were to be used. To demonstrate zonisamide's effectiveness in a representative Veteran sample, the investigators will include Veterans with co-morbid mood and anxiety disorders.

The investigators also plan to explore the interaction between genotype and medication on drinking outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Female/male veterans aged 21-70 years
* Regular heavy drinkers as defined by averaging 2 heavy drinking days per week over 90 days baseline pre-treatment timeline follow-back (TLFB), and current alcohol dependence diagnosis by the Diagnostic and Statistical Manual IV Text Revision (DSM-IV-TR) that recognize a need to reduce or stop drinking (Note: heavy drinking days will be defined as follows; for men greater than or equal to 5 drinks in a day and for women greater than or equal to 4 drinks in a day)
* Women of child-bearing potential (i.e., no hysterectomy, bilateral oophorectomy, or tubal ligation or <2 years postmenopausal), must be non-lactating, practicing a reliable method of birth control, and have a negative serum pregnancy test prior to initiation of treatment;
* Willingness to provide signed, informed consent to participate in the study

Exclusion Criteria:

* A current, clinically significant physical disease or abnormality (i.e., neurologic, renal, rheumatologic, gastrointestinal, hematologic, pulmonary, endocrine, cardiovascular, hepatic, or autoimmune disease that, in the context of the study would represent a risk to the subject, or significant laboratory abnormalities such as hepatic aminotransferase levels [i.e., aspartate aminotransferase (AST) and alanine aminotransferase (ALT)] greater than 300% of the upper limit of normal or direct bilirubin levels >150% of the upper limit of normal) on the basis of medical history, physical examination, or routine laboratory evaluation. Other specific exclusionary disorders include;
* History of renal calculi or renal failure; a significant indication of renal compromise will be defined by an elevation of serum creatinine above the investigators' laboratory's limit of normal, or a known history of renal failure or chronic renal disease, or any current or chronic disease that could reasonably be expected to result in renal failure
* History of hypersensitivity to zonisamide or any sulfonamide, Stevens-Johnson Syndrome, penicillin allergy, or history of any severe drug allergic reaction;
* History of systemic autoimmune disease such as lupus erythematosis, fibromyalgia, or rheumatoid arthritis;
* Current blood dyscrasia or a history of such, with the exception of a past history of iron deficiency anemia
* History of seizure disorder
* Use of any of a number of medications that might prominently influence drinking patterns or cause risk of harm or injury (e.g., topiramate, disulfiram, naltrexone, acetazolamide, stimulants such as amphetamine, or tramadol;
* Schizophrenia, bipolar disorder, posttraumatic stress disorder (PTSD), or substantial suicide or violence risk (i.e., can't be managed safely in the outpatient setting) on the basis of history or psychiatric examination; j) currently dependent on opioids or benzodiazepines or other sedatives
* Considered by the investigators to be clinically inappropriate for study participation or have participated in another pharmacotherapy study in the past thirty days
* Subjects with prominent signs of physical dependence, and/or medical comorbidities such that study physicians feel they should consider immediate detoxification, and referred for medical detoxification in a normal treatment setting

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert J Arias, MD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (1):
- VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomization was conducted by the pharmacy using a 1:1 randomization in blocks of 4 and stratified by site.
Groups:
- Zonisamide: Participants received zonisamide titrated to a target dose of 500mg orally, daily, double-blind (Titration of dose to 500mg oral, daily, over 8 weeks, then 7 weeks of treatment at that dose). Subjects may increase their dose to 600mg daily during the target treatment period if it is thought to be beneficial.
  Zonisamide: Titration of dose to 500mg oral, daily, over 8 weeks, then 7 weeks of treatment at that dose
- Placebo: Participants received placebo pills that are made to match the zonisamide medication (via over-encapsulation, double-blind, subjects will receive same number of capsules as the active medication group) Placebo: Placebo
Period: Overall Study
Arm/Group | Zonisamide | Placebo
Started | 46 | 46
Completed | 22 | 27
Not Completed | 24 | 19

BASELINE CHARACTERISTICS:
Population: All available data was utilized in the analysis using mixed models
Groups:
- Zonisamide; Placebo: Men or women veterans, ages 21-70, met Diagnostic and Statistical Manual IV Text Revision (DSM-IV) criteria for current Alcohol Dependence (AD) (determined by structured clinical interview)
- Total: Total of all reporting groups
Arm/Group | Zonisamide | Placebo | Total
Number analyzed (Participants) | 43 | 45 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (11.7) | 51.8 (10.8) | 50.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All available data was utilized in the analysis using mixed models
  Participants
    number analyzed (Participants) | 42 | 44 | 86
    Female | 3 | 2 | 5
    Male | 39 | 42 | 81
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 31 | 31 | 62
  African American | 11 | 11 | 22
  Other | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Drinks Per Week
Description: Difference between groups in the number of total standard drinks per week over 8 weeks (weeks 9-16, the weeks on the target dose) performed using a mixed models longitudinal analysis.
Time Frame: over 8 weeks (weeks 9-16)
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: Number of total drinks
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 43 | 46
Number of total drinks
  Week 9 | 17.8 (7.6) | 8.1 (7.5)
  Week 10 | 12.2 (4.6) | 8.8 (4.5)
  Week 11 | 15.9 (5.6) | 3.6 (5.5)
  Week 12 | 10.3 (3.6) | 6.2 (3.6)
  Week 13 | 9.4 (6.9) | 12.5 (6.3)
  Week 14 | 9.9 (3.4) | 4.3 (3.1)
  Week 15 | 13.7 (4.1) | 3.3 (3.7)
  Week 16 | 11.1 (5.1) | 8.7 (4.3)

2. Secondary Outcome: Percentage of Subjects With No Heavy Drinking Days (PSNHDD)
Description: Percentage of Subjects with No Heavy Drinking Days (PSNHDD) The PSNHDD can be derived from each subject's timeline follow back (TLFB) data.
Time Frame: Baseline
Population: All available data was utilized in the analysis using mixed models
Measure: Count of Participants; unit: Participants
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 43 | 46
Participants
  Participants with No Heavy Drinking Days | 16 | 28
  Participants with Heavy Drinking Day | 27 | 18

3. Secondary Outcome: Gamma Glutamyl Transferase (GGT)
Description: Difference between groups on change in levels of Gamma glutamyl transferase (GGT) over time from baseline to endpoint, which will include several interim data points. This will analyzed with a mixed models longitudinal analysis (repeated measures). Normal range for GGT levels are 10 U/L - 65 U/L - above 65 U/L above 65 U/L is considered a high GGT level
Time Frame: Baseline, Week 4, 8 and 16
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: Units/Liter (U/L)
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 43 | 46
Units/Liter (U/L)
  Baseline | 76.0 (12.7) | 78.2 (12.2)
  Week 4 | 63.4 (8.8) | 50.0 (8.7)
  Week 8 | 61.40 (8.8) | 45.5 (8.7)
  Week 16 | 62.8 (10.2) | 46.4 (9.9)

4. Secondary Outcome: Number of Heavy Drinking Days Per Week
Description: The difference in the number of heavy drinking days per week compared between groups (zonisamide and placebo) during the time spent on the target dose of the medication. Performed using a mixed models longitudinal analysis (repeated measures).
Time Frame: over 16 weeks (weeks 1-16)
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: Number of heavy drinking days
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 43 | 46
Number of heavy drinking days
  Week 1 | 1.1 (0.3) | 0.6 (0.3)
  Week 2 | 0.9 (0.3) | 0.9 (0.3)
  Week 3 | 0.8 (0.3) | 0.8 (0.3)
  Week 4 | 1.1 (0.3) | 0.3 (0.3)
  Week 5 | 0.8 (0.3) | 0.5 (0.3)
  Week 6 | 0.8 (0.3) | 0.6 (0.3)
  Week 7 | 0.8 (0.3) | 0.6 (0.3)
  Weel 8 | 1.0 (0.3) | 0.5 (0.3)
  Week 9 | 1.0 (0.3) | 0.5 (0.3)
  Week 10 | 1.0 (0.3) | 0.5 (0.3)
  Week 11 | 0.8 (0.3) | 0.4 (0.3)
  Week 12 | 0.8 (0.3) | 0.5 (0.3)
  Week 13 | 0.7 (0.3) | 0.3 (0.2)
  Week 14 | 0.9 (0.3) | 0.2 (0.3)
  Week 15 | 0.8 (0.3) | 0.5 (0.3)
  Week 16 | 11.4 (3.1) | 6.5 (3.0)

5. Secondary Outcome: Alcohol Urge Questionnaire Score (AUQ)
Description: This is the change in AUQ scores (urge to drink) measured weekly compared between groups using repeated measures. The AUQ is a 8 item participant rated questionnaire. Participants indicate how much they agree or disagree with the statements by selecting one number, 1 strongly disagree through 7 strongly agree. Participants can scores between 8 (lowest) - 56 (highest), the higher the score the more urge to drink.
Time Frame: over 16 weeks (weeks 1-16)
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 43 | 46
units on a scale
  Baseline | 17.1 (1.2) | 14.8 (1.2)
  Week 1 | 13.3 (1.1) | 12.7 (1.0)
  Week 2 | 14.0 (1.2) | 11.8 (1.2)
  Week 3 | 14.7 (1.1) | 10.7 (1.1)
  Week 4 | 13.5 (1.0) | 10.7 (1.0)
  Week 5 | 13.6 (1.1) | 10.7 (1.1)
  Week 6 | 12.3 (1.2) | 10.7 (1.2)
  Week 7 | 12.7 (1.1) | 12.1 (1.1)
  Week 8 | 12.4 (1.1) | 11.3 (1.1)
  Week 9 | 13.4 (1.2) | 11.0 (1.2)
  Week 10 | 11.9 (1.0) | 10.7 (0.9)
  Week 11 | 10.9 (0.8) | 10.9 (0.8)
  Week 12 | 11.7 (1.0) | 10.3 (0.9)
  Week 13 | 10.3 (0.8) | 10.3 (0.8)
  Week 14 | 11.8 (1.2) | 9.8 (1.2)
  Week 15 | 10.8 (0.8) | 9.7 (0.8)
  Week 16 | 12.0 (1.0) | 9.8 (1.0)

6. Secondary Outcome: Change in Quality of Life
Description: Change in quality of life scores measured by the Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q). The Q-LES-Q is a 16 item participant rated questionnaire. Participants indicate how they are feeling over the 16 item from Very poor (1), Poor (2), Fair (3), Good (4), and Very Good (5). Participants can scores between 14 (lowest) - 70 (highest) the higher the score more satisfied with quality of life.
Time Frame: Over 16 weeks (Baseline and 16 weeks)
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 43 | 46
units on a scale
  Baseline | 56.9 (2.7) | 55.8 (2.6)
  Week 16 | 73.3 (3.5) | 72.9 (3.1)

7. Secondary Outcome: Level of Alcohol-related Problems (SIP)
Description: Change in level of alcohol-related problems measured by the Short Index of Problems (SIP). The SIP is a 15 item participant rated questionnaire. Participants rate the number of events that drinkers sometimes experience. Participants indicate how often each of the items has happened. They are scored by selecting one number, 0 Never; 1 Once or a few times; 2 Once or twice a week; 3 Daily or almost daily. Participants can scores between 0 (lowest) - 45 (highest) - the higher score the more drinking problems.
Time Frame: over 16 weeks (Baseline and Week 16)
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 43 | 46
units on a scale
  Baseline | 4.8 (0.4) | 5.3 (0.4)
  Week 16 | 1.2 (0.5) | 1.9 (0.5)

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: Adverse events were collected with a questionnaire of side effects at appointments over the 16 week period.
Arm/Group | Zonisamide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/46
Serious Adverse Events (participants affected / at risk) | 4/46 | 0/46
Other Adverse Events (participants affected / at risk) | 2/46 | 6/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zonisamide (N=46) | Placebo (N=46)
Suicidal Ideation (Psychiatric disorders) | 3 (3) | 0 (0) — Hospitalized for detox and suicidal ideation
Homicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0) — hospitalized
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zonisamide (N=46) | Placebo (N=46)
Alcohol detoxification (Psychiatric disorders) | 2 (2) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/31/NCT02368431/Prot_SAP_000.pdf